CLINICAL TRIAL: NCT04873882
Title: Waveform and Spectral Characteristics of Perioperative Wheezing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Allison Bechtel, MD, Assistant Professor of Anesthesiology, University of Virginia
Other Study IDs: 21550
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Sounds; Thoracic Surgery
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Acoustic ventilation — 1. Placement and removal of the esophageal stethoscope
  2. Connection of a microphone to the esophageal stethoscope outside of and removed from the patient's body at the location on the figure above "Connection fo monaural earpiece."
  3. Digital breath sound real-time monitoring will be collected as .wav files from the device with no identifiable elements and the data from the device will be downloaded onto a desktop and we will keep and store the data on a secure departmental server.
  4. Additional monitoring schedule includes evaluation of breath sounds with a conventional stethoscope every 30 minutes intraoperatively, at the start of one-lung ventilation, at the return to two-lung ventilation and prior to extubation and during any changes on the digital breath sounds recording monitor.

SUMMARY:
With the aid of computerized sound analysis, digital acoustic monitoring could provide a more sensitive, specific, and quantifiable indicator for perioperative respiratory abnormalities including wheezing. It is probable that the digital stethoscope has utility in the detection, monitoring, and resolution following treatment of acoustic changes characteristic of turbulent respiratory gas flow due to wheezing and/or the incomplete resolution of atelectasis following the re-initiation of ventilation in a collapsed lung.

DETAILED DESCRIPTION:
Anesthesiologists still rely on use of a conventional stethoscope to detect abnormal breath sounds during and after surgery - this process is labor intensive, intermittent, relies on human experience and thus is highly subjective. In fact, even for the most basic assessments, e.g. endobronchial intubation, human auscultation is unreliable.1 Digital stethoscopes are able to both amplify and digitize airway sounds and also provide a mechanism to record and analyze them for features undetectable by a human. Several small, pilot studies have shown that acoustic waveforms from the lungs produce characteristic spectral patterns in specific pulmonary pathophysiologic states. At this time, there are no studies that examine the acoustic patterns specific to perioperative wheezing or lung re-expansion. With the aid of computerized sound analysis, digital acoustic monitoring could provide a more sensitive, specific, and quantifiable indicator for perioperative respiratory abnormalities including wheezing. It is probable that the digital stethoscope has utility in the detection and monitoring of acoustic changes characteristic of turbulent respiratory gas flow due to wheezing and/or the incomplete resolution of atelectasis following the re-initiation of ventilation in a collapsed lung. In addition, treatment of perioperative wheezing with an inhaled bronchodilator may lead to resolution of wheezing and this response to treatment may also be monitored using waveform and spectral characteristics of the acoustic patterns from the digital stethoscope.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for either:

1. open thoracic or video-assisted thoracoscopic surgery under general anesthesia requiring one-lung ventilation
2. abdominal surgery with a known history of chronic obstructive pulmonary disease (as documented in the electronic medical record)

Exclusion Criteria:

* Emergency surgery
* surgery requiring the use of transesophageal echocardiography
* refusal of informed consent
* pregnancy
* esophageal surgery
* lung transplantation
* contraindications for placement of esophageal stethoscope including esophageal varices strictures, motility disorders, diverticula or a history of prior esophageal injury or surgery
* age less than 18 years old
* prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing the following procedures:
  1. open thoracic or video-assisted thoracoscopic surgery under general anesthesia requiring one-lung ventilation
  2. abdominal surgery with a known history of chronic obstructive pulmonary disease (as documented in the electronic medical record)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-08-27 (Estimated); Study Completion 2021-08-27 (Estimated)

PRIMARY OUTCOMES:
Spectral Waveform Analysis to discriminate between wheezing and not wheezing based on specific frequency bands | Duration of the operation while the esophageal stethoscope is in place, an average of 3 hours
  Comparison of the spectral waveforms to determine the specific frequency bands associated with wheezing and non-wheezing

SECONDARY OUTCOMES:
Spectral waveform analysis associated with ventilatory parameters | Duration of the operation while the esophageal stethoscope is in place, an average of 3 hours
  Ventilatory parameters including respiratory rate, tidal volume, and airway pressures that were recorded during the case will be compared with the spectral waveforms to determine the specific frequency bands associated with ventilatory parameters during one-lung ventilation and two-lung ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No